CLINICAL TRIAL: NCT03005587
Title: Impact of Acute Decompensation in Patients of Cirrhosis With or Without Prior Decompensation - A Prospective Observational Study.
Brief Title: Impact of Acute Decompensation in Patients of Cirrhosis With or Without Prior Decompensation
Status: Withdrawn | Type: Observational
Why Stopped: Lack of Funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-Cirrhosis-06
Record Dates: First submitted 2016-12-23; First posted 2016-12-29 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Acute Decompensation in Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cirrhotics with no previous decompensation
- Cirrhotics with previous one or more than one decompensation

SUMMARY:
This a prospective observational study in Chronic Liver Disease patients admitted or seen in OPD, Department of Hepatology, Institute of Liver and Biliary Sciences, India. The study will be conducted in a period of three months starting September 2016 in sample size of 80 . A detailed proforma including history and examination and routine blood investigations will be noted. The patients will undergo close follow up at 0, 7, 15, 30, 45, 60, 90 days and similar activities will be repeated at every visit.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis with decompensation in a period of 3 months in form of ascites, jaundice, Hepatic Encephalopathy, Acute Variceal bleed irrespective of prior decompensation.
2. Age 18-70 years
3. Valid consent

Exclusion Criteria:

1. HepatoCellular Carcinoma
2. Admitted and survival less than 48 hrs
3. Pregnant
4. Acute Liver Failure
5. Post transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic liver disease patients admitted or seen in Out Patient Department, Department of Hepatology, Institute of Liver & Biliary Sciences, India.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-12-31 (Estimated); Primary Completion 2017-03-01 (Estimated); Study Completion 2017-03-01 (Estimated)

PRIMARY OUTCOMES:
Spontaneous recovery or liver transplant or death in both groups | 90 days

SECONDARY OUTCOMES:
Cause of acute decompensation | 3 months
Severity and duration of prior as well as present decompensation | 3 months
Improvement in severity assessment Indices Model for End Stage Liver Disease in both groups. | 3 months
Causes of death in both groups | 3 months
Profile of patient undergone transplant in both groups | 3 months
Sepsis in both groups | 3 months
Systemic Inflammatory Response Syndrome in both groups | 3 months
Improvement in severity assessment Indices Child Pugh Turcotte in both groups. | 3 months
Improvement in severity assessment Indices Sequential Organ Failure Assessment in both groups | 3 months
Improvement in severity assessment Indices Acute Physiology and Chronic Health Evaluation II in both groups | 3 months
Improvement in severity assessment Indices CLIF score in both groups | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences., New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No